CLINICAL TRIAL: NCT00245726
Title: Lower Extremity Cycling With Functional Electrical Stimulation to Improve the Health and Fitness of Children With Spinal Cord Injuries
Brief Title: Functional Electrical Stimulation (FES) Cycling for Children With Spinal Cord Injuries (SCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Richard T. Lauer, Shriners Hospitals for Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHC-8540
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Passive (Motor Assist) Cycle
  Interventions: Device: Passive (Motor Assist) Cycle
- 2 (Active Comparator)
  Interventions: Device: ES therapy
- 3 (Experimental)
  Interventions: Device: FES Cycle

INTERVENTIONS:
Device: FES Cycle — Subjects will use electrical stimulation of the leg muscles to pedal a cycle for 1 hour / 3x week
  Arms: 3
Device: ES therapy — Subjects will electrically stimulate the leg muscles for 1 hour/ 3x week
  Arms: 2
Device: Passive (Motor Assist) Cycle — Subjects will use a cycle that moves the legs for 1 hour/3x per week
  Arms: 1

SUMMARY:
The overall objective of this research project is to examine the clinical efficacy of lower extremity cycling with functional electrical stimulation to improve the health and fitness of children with spinal cord injuries (SCI). To achieve this goal, a controlled, randomized study will be conducted with thirty children who have sustained a spinal cord injury. The children in the study will be assigned to one of three groups: those receiving functional electrical stimulation (FES) leg cycling exercise, those receiving passive leg cycling, and a non-cycling control group receiving electrical stimulation therapy to generate muscle contractions in the lower extremity. All three groups will be balanced as to the amount of time they receive the specific therapy. All therapies, after initial assessment, will be conducted at home in order to foster changes in lifestyle that may prove to be essential for improved quality of life.

The specific aims of this proposal are delineated below:

Aim 1: To assess, by means of a randomized controlled study design, the ability of FES cycling to improve the cardiovascular and musculoskeletal systems of ten children with a spinal cord injury, as compared to ten children undergoing passive leg cycling exercise and ten children receiving electrical stimulation therapy alone.

Aim 2: To determine, by means of a randomized controlled study design, the feasibility of using FES leg cycling exercise to provide long-term health benefits and improve the neurologic status of ten children with a spinal cord injury, as compared to ten children undergoing passive leg cycling exercise and ten children receiving electrical stimulation therapy alone.

DETAILED DESCRIPTION:
This is a controlled, randomized pretest/posttest study design in which three conditions will be compared: FES leg cycling exercise, passive leg cycling exercise, and a control group receiving electrical stimulation therapy. Randomization of the subjects into the three groups will be coordinated across the two sites. All other variables will be controlled to the extent possible. All children in this study will continue to receive standard therapy at the level established by the therapist working with the child. This includes passive stretching of the lower extremities and the use of standing frames. Medications will also remain unaltered throughout the study, unless changes in body mass or other physical conditions unrelated to the study (i.e. growth) warrant modification. All exercise sessions, after the initial one or two-week assessment, will be conducted at home.

Electrical activation of the muscles in this study will be achieved through the use of surface mounted electrodes. The muscle groups that will be electrically activated in this study are the quadriceps, the hamstrings, and the gluteal muscles bilaterally. This is based upon the previous FES cycling studies conducted in the adult population. The appropriate stimulation levels for each muscle will be determined for each subject.

All subjects in the three study groups, in addition to participation in this study, will receive standard therapy at home. For all of the children, this will include passive range of motion stretching three times each week. Ideally, stretching will be done before cycling or electrical stimulation therapy to act as a "warm-up" period before the more involved therapies are performed. For the children with sustained tetraplegia participating in this study, standard therapy will also involve standing three times each week, either with braces or the use of a standing frame.

FES Cycling Group The FES cycling group will be asked to participate in additional therapy involving cycling for thirty minutes, three times a week. All cycling movements will be accomplished with electrical activation of the leg muscles. The first one to two weeks will be conducted on-site to monitor the subjects' reaction to exercise, after which therapy sessions will continue at home. The goal will be achieving thirty minutes of continuous cycling at 50 rev•min-1 with zero power output. Until subjects reach this point, the cycling session will be divided into five to ten minute-long sets, separated by five-minute rest breaks. Each subject, however, will complete a total of thirty minutes of cycling at the set speed. Once subjects reach this point, the power output requirements will be increased. From the zero point, the power requirement for the first session will be increased by one watt (W). If the subject can cycle continuously for 30 minutes, the next session the power output requirement will be increased by one watt. If the subject cannot pedal for a full 30 minutes, the power requirement will be maintained at this higher level until 30 minutes of continuous cycling can be achieved. The power requirement will then be increased by one watt on the next session. Increases will continue in this manner until the end of the protocol, or until the maximum power output of 50 watts, has been reached.

Passive Cycling Group The passive cycling group will be asked to participate in additional therapy that will also involve cycling for thirty minutes, three times a week. However, the motor in the bicycle will provide all cycling movements. The first one to two weeks will be conducted on-site under the observation of the investigators, after which time therapy sessions will continue at home. The initial sessions will be used to determine whether the subject can tolerate the exercise, and to build fatigue resistance. The goal will be to achieve thirty minutes of continuous cycling at 50 rev•min-1 with zero power output. Once subjects can cycle for thirty minutes continuously, the subjects will continue at this level until the completion of the protocol.

Electrical Stimulation Therapy Group Subjects in the control group will maintain their standard therapy, in addition to receiving additional electrical stimulation therapy of the quadriceps and hamstring muscles for a period of 30 minutes, three times per week. The children in this group will act as a control group for the comparison of additional therapy time involving cycling, as compared to additional therapy time only. Electrical stimulation was selected as the additional therapy of choice since specific health and physiologic benefits have already been reported by this group of investigators and could thus be seen as comparable to cycling. Stimulation of the muscles will be accomplished using a portable, 2-channel surface stimulation unit (Empi, St. Paul Minnesota) instead of the ExoStim Unit. The hamstrings and quadriceps will be activated bilaterally for 15 minutes each at a level that produces a strong muscle contraction. This will be accomplished while the subjects are resting in the supine position, working against zero resistance. Attempts will also be made to incorporate the gluteal muscles into the electrical stimulation protocol, but the sessions will not exceed the thirty-minute time period.

ELIGIBILITY:
Inclusion Criteria:

1. Satisfactory general health
2. Twelve months post injury to allow for plateau in neurology function, bowel patterns, and cardiovascular patterns
3. Cervical (tetraplegia) or thoracic (paraplegia) level spinal cord injury (ASIA A and ASIA B classifications)
4. Intact lower motor neurons of the targeted lower extremity muscles
5. Skeletally immature (5 to 15 years of age)
6. Ability to maintain an upright position with minimal support
7. Adequate time available for trial participation (12 months)

Exclusion Criteria:

1. Conditions (e.g. arthritis) requiring chronic steroid treatment
2. Symptomatic or known cardiac disease
3. Presence of a seizure disorder
4. Pulmonary disease limiting exercise tolerance
5. Conflicting implanted devices which may be adversely affected by the electrical stimulation (any implanted medical device, including a cardiac pacemaker or electronic Baclofen pump)
6. History of lower limb stress fractures
7. Severe spasticity in legs - score of ³ 4 on the Modified Ashworth scale
8. Presence of a Grade 2 or higher pressure area on the legs, buttocks, or trunk
9. Severely limited range of joint motion/irreversible muscle contractures
10. Ossification of joints in the lower limbs
11. Hip instability / dislocation
12. History of uncontrolled autonomic dysreflexia
13. Previous participant in electrical stimulation or activity based therapy (i.e. cycling, treadmill training) within 3 months of enrollment
14. Small size of the subject limiting the ability to be safely positioned on the bicycle

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Muscle Cross Sectional Area | 6 months
ES Muscle Strength | 12 months
Bone Mineral Density of Hip and Knee | 12 months
Cholesterol | 12 months
White Blood Cell Count | 12 months
Peak Resistive Force | 12 months
Ashworth Scale | 12 motnhs
Spasm Scale | 12 months
Quality of Life (PedsQL) | 12 months
ASIA assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lauer, PhD, Principal Investigator — Shriners Hospitals for Children; John W McDonald, MD, PhD, Principal Investigator — Kennedy Kreiger Institute
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Shriners Hospitals for Children, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Johnston TE, Modlesky CM, Betz RR, Lauer RT. Muscle changes following cycling and/or electrical stimulation in pediatric spinal cord injury. Arch Phys Med Rehabil. 2011 Dec;92(12):1937-43. doi: 10.1016/j.apmr.2011.06.031. PMID 22133240
- [Derived] Johnston TE, Smith BT, Mulcahey MJ, Betz RR, Lauer RT. A randomized controlled trial on the effects of cycling with and without electrical stimulation on cardiorespiratory and vascular health in children with spinal cord injury. Arch Phys Med Rehabil. 2009 Aug;90(8):1379-88. doi: 10.1016/j.apmr.2009.02.018. PMID 19651272